CLINICAL TRIAL: NCT00071006
Title: Phase 2 Study Of AG-013736 In Patients With Poor Prognosis Acute Myeloid Leukemia (AML) Or Myelodysplastic Syndrome (MDS)
Brief Title: AG-013736 (Axitinib) In Patients With Poor Prognosis Acute Myeloid Leukemia (AML) Or Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061013
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Results first posted 2012-03-19 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-05

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study (Experimental)
  Interventions: Drug: AG-013736 (Axitinib)

INTERVENTIONS:
Drug: AG-013736 (Axitinib) — patients were treated with axitinib at starting dose of 5 mg BID continuous dosing.

SUMMARY:
The study tests the safety and efficacy of axitinib in patients who have the hematologic disease of Acute Myeloid Leukemia or Myelodysplastic Syndrome. The study tests patients who have poor prognosis before entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Poor prognosis AML or MDS
* Histological confirmation of diagnosis
* White blood cell count less than or equal to 30,000/mm3
* Adequate hepatic and renal function documented within 14 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* No evidence of preexisting uncontrolled hypertension
* Not a suitable candidate for chemotherapy
* No prior systemic chemotherapy treatment for AML or MDS or treatment with an anti-angiogenesis agent

Exclusion Criteria:

* Patients must not have exclusion criteria.
* Candidate for chemotherapy
* Patients with AML M3 (acute promyelocytic leukemia)
* Conditions that might confound the evaluation of safety or efficacy or increase patient risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-09; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Houston, Texas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061013&StudyName=AG-013736%20%28Axitinib%29%20In%20Patients%20With%20Poor%20Prognosis%20Acute%20Myeloid%20Leukemia%20%28AML%29%20Or%20Myelodysplastic%20Syndrome%20%28MDS%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 milligram (mg) twice daily (BID) continuously. Treatment was administered continuously until progression, relapse, failure, or disease transformation or toxicity occurred.
Period: Overall Study
Arm/Group | Axitinib
Started | 12
Completed | 0
Not Completed | 12
Not completed — Lack of Efficacy | 7
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: Years] | 77.42 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Participants with OR based on a assessment of confirmed complete remission (CR) or partial remission (PR) according to Cheson criteria for Acute myeloid leukemia (AML) and Myelodysplastic syndrome (MDS). CR: those with > 20% cellularity of bone marrow biopsy, no presence of extramedullary leukemia for AML, <5 % myeloblast cells for bone marrow with peripheral blood value lasting at least 1 month and 2 months for AML and MDS respectively. PR : those with all criteria for CR except 5-25 % blasts in bone marrow and at least 50% decrease in blast over pretreatment for AML and MDS respectively.
Time Frame: Baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 4 weeks up to 35 weeks
Population: Study Population included all participants who received at least 1 dose of study medication and had a baseline assessment of disease.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 12
Percentage of participants | 0 [0 to 0.265]

2. Secondary Outcome: Percentage of Participants With Hematologic Improvement (HI)
Description: HI was described by the number of individual and positively affected cell lines (Erythroid response, Platelet response, Neutrophil response). Improvements must last at least 2 months.
Time Frame: Baseline, Week 2 thereafter every 4 weeks up to 35 weeks and follow up (at least 30 days after last dose)
Population: Analysis for this particular endpoint was not conducted due to lack of efficacy.
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1). DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: First documentation of objective response until objective disease progression or discontinuation from the study due to any cause assessed every 4 weeks up to 35 weeks
Population: Analysis for this particular endpoint was not conducted due to lack of efficacy.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Bone Marrow Micro Vessel Density (MVD)
Description: Bone marrow MVD in tumors is a measure of angiogenesis and a prognostic indicator that correlates with an increased risk of metastasis in various cancers and with overall and relapse free survival in participants with AML or MDS. Bone marrow biopsies and bone marrow clot samples were assessed for MVD (cluster of differentiation 31 [CD31] staining).
Time Frame: Day 1, Week 2 thereafter every 4 weeks up to 35 weeks
Population: Data was not summarized for this particular endpoint due to lack of efficacy.
Measure: Mean (Standard Deviation); unit: vessels/square millimeter (mm^2)
Arm/Group | Axitinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Vascular Endothelial Growth Factor Receptor 1 (VEGFR-1) and VEFGR Receptor 2 (VEGFR-2) Phosphorylation
Description: Vascular endothelial growth factor (VEGF) promotes cancer progression by inducing angiogenesis via VEGF receptors, signals directly through receptors VEGFR-1 and VEGFR-2. Change in biomarkers related to VEGFR signal transduction pathways after axitinib treatment was assessed. Mononuclear (MNC) cell VEGF receptor expression and phosphorylation was assessed by in situ western blot analysis. VEGFR-1 and VEGFR-2 evaluations were performed using samples from peripheral blood plasma, bone marrow aspirate, bone marrow (Core) biopsy and bone marrow clot.
Time Frame: Day 1, Week 2 thereafter every 4 weeks up to 35 weeks and follow up (at least 30 days after last dose)
Population: Data was not summarized for this particular endpoint due to lack of efficacy.
Measure: Mean (Standard Deviation); unit: picograms (pg)/mL
Arm/Group | Axitinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Plasma Vascular Endothelial Growth Factor (VEGF) Concentration
Description: VEGF promotes cancer progression by inducing angiogenesis via VEGF receptors, signals directly through receptors VEGFR-1 and VEGFR-2. Change in biomarkers related to VEGFR signal transduction pathways after axitinib treatment was assessed. Plasma VEGF concentration evaluations were performed using samples from peripheral blood plasma, bone marrow aspirate, bone marrow (Core) biopsy and bone marrow clot.
Time Frame: Day 1, Week 2 thereafter every 4 weeks up to 35 weeks and follow up (at least 30 days after last dose)
Population: Data was not summarized for this particular endpoint due to lack of efficacy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Axitinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Population Pharmacokinetics of Axitinib (AG-013736)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Day 1 (pre-dose) and every 4 weeks up to 35 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: ng/mL

8. Secondary Outcome: Overall Survival (OS)
Description: Time in days from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1). Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death). For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline to death due to any cause or at least every 3 months after discontinuation of study treatment
Population: Analysis for this particular endpoint was not conducted due to lack of efficacy.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood pressure increased (Investigations) | 2
Cardiac murmur (Investigations) | 1
Platelet count decreased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear disorder (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Dry eye (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oral disorder (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 4
Tongue disorder (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 3
Chills (General disorders) | 3
Fatigue (General disorders) | 9
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 4
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Laryngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood pressure increased (Investigations) | 2
Carbon dioxide increased (Investigations) | 1
Cardiac murmur (Investigations) | 1
Carotid bruit (Investigations) | 1
Weight decreased (Investigations) | 2
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 1
Muscle contractions involuntary (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.